CLINICAL TRIAL: NCT00868452
Title: A Randomized, 6-Week, Double-Blind, Placebo- Controlled, Flexible-Dose, Parallel-Group Study of Lurasidone Adjunctive to Lithium or Divalproex for the Treatment of Bipolar I Depression
Brief Title: Lurasidone - A 6-week Study of Patients With Bipolar I Depression (Add-on)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1050235; EUDRACT No. 2008-007482-23
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar Depression
Keywords: Bipolar I; Latuda; Lurasidone
MeSH Terms: conditions — Bipolar Disorder | interventions — Lurasidone Hydrochloride; Lithium; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lurasidone (Experimental)
  Interventions: Drug: lurasidone + (lithium or divalproex)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo + (lithium or divalproex)

INTERVENTIONS:
Drug: lurasidone + (lithium or divalproex) — lurasidone 20 mg/day for Days 1-2-3, 40 mg/day for Days 4-5-6, and 60 mg/day on Day 7.
  Arms: Lurasidone
Drug: Placebo + (lithium or divalproex) — 20 mg/day for Days 1-2-3, 40 mg/day for Days 4-5-6, and 60 mg/day on Day 7
  Arms: Placebo

SUMMARY:
This clinical study is designed to test the hypothesis that lurasidone is effective, tolerable, and safe when added to treatment with lithium or Divalproex for the treatment of patients with bipolar I depression.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with bipolar I disorder, most resent episode depressed
* Subject must have a lifetime history of at least one bipolar manic or mixed episode
* Subject must be taking lithium or divalproex at least 28 days prior to screening

Exclusion Criteria:

* History of nonresponse to an adequate (6-week) trial of three or more antidepressants (with or without mood stabilizers) during the current episode
* Subject has been hospitalized for a manic or mixed episode within 60 days prior to randomization
* Imminent risk of suicide or injury to self, others, or property

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (71):
- United States (27):
  - Woodland International Research Inc., Little Rock, Arkansas
  - South Coast Clinical Trials, Inc., Anaheim, California
  - Catalina Research Institute, Chino, California
  - Synergy Escondido, Escondido, California
  - Collaborative Neuroscience Network Inc.,12772 Valley View Street, Garden Grove, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California at Irvine Medical Center, Orange, California
  - CNRI - Los Angeles LLC,8309 Telegraph Road, Pico Rivera, California
  - CNRI - San Diego, LLC, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Depression and Anxiety Disorders Research Institue, Tampa, Florida
  - American Medical Research Inc.,1200 Harger Road Suite 415, Oak Brook, Illinois
  - American Medical Research, Inc., 1200 Harger Road Suite 415, Oak Brook, Illinois
  - J. Gary Booker, MD, Shreveport, Louisiana
  - Sheppard Pratt Health System,6501 North Charles Street, Baltimore, Maryland
  - Capital Clinical Research,5515 Security Lane, Suite 525, Rockville, Maryland
  - Midwest Research Group, Saint Charles, Missouri
  - Albuquerque Neuroscience Inc.,101 Hospital Loop, Suite 209, Albuquerque, New Mexico
  - Lake Charles Clinical Trials LLC,700 Spring Forest Road, Raleigh, North Carolina
  - Richard H. Weisler , M.D., PA.,& Associates, 700 Spring Forest Road, Suite 125, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Mood Disorders Program-UHCMC, Cleveland, Ohio
  - MetroHealth System, Cleveland, Ohio
  - Midwest Clinical research Center, One Elizabeth Place, Suite G-3, Dayton, Ohio
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, LLC., 4200 Marathon Blvd., Suite 200, Austin, Texas
- Czechia (5):
  - Psychiatricka ambulance, Brno - Mesto
  - BIALBI s.r.o. Psychiatricke oddeleni, Litoměřice
  - Clintrial, s.r.o., Prague
  - Medical Services Prague s.r.o., Prague
  - Psychiatricka ambulance Prosek, Prague
- France (2):
  - Hopital Caremeau, Service de Psychiatrie A, Nîmes
  - Zans Ritter, Marcel, Orvault
- Jana Thomsen, Berlin BE, Germany
- India (11):
  - SV Medical College, Tirupati, Andh Prad
  - Vijayawada Institute of Mental Health and Neurosciences, Psychiatry, Vijaywada, Andh Prad
  - Samvedna Hospitals, Ahmedabad, Gujarat
  - Sheth Vadilal Sarabhai General Hospital, Ahmedabad, Gujarat
  - Mental Illness Treatment Rehabilitation Foundation (MITR), Ahmedabad, Gujarat
  - Shree Hatkesh Health Foundation, Jūnāgadh, Gujarat
  - Spandana Nursing Home, Bangalore, Karna
  - Sujata Birla Hospital & Research Centre, Nashik, Mahara
  - Cosmos Hospitals-Delhi Psychiatry Center-Dept. of Psychiatry, Delhi, National Capital Territory of Delhi
  - R.K. Yadav Memorial Mental Health & De-Addiction Hospital, Jaipur, Rajasthan
  - Manobal Med. Research Centre, Lucknow, Uttar Prad
- Poland (3):
  - ZOZ Poradnia Zdrowia Psychicznego, Chełmno
  - Praktyka Lekarska Sensorium S.M.O., Skorzewo
  - Wojewodzki Szpital Brodnowski SP ZOZ, Warsaw
- Romania (6):
  - Spitalul Clinic de Urgenta Militar Central "Prof. Dr. Carol" Psihiatrie, Bucharest
  - Spitalul Clinic de Psihaiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova
  - Spitalul Clinic de Neurologie si Psihiatrie Oradea, Oradea
  - Spitalul Judetean de Urgenta Pitesti Sectia de Psihiatric, Piteşti
- Russia (6):
  - Russian State Medical University, Moscow
  - Moscow Medical Academy named I.M. Sechenov, Moscow
  - City Psychiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - Bekhterev Scientific Research Psychoneurological Institute, Saint Petersburg
  - Psychoneurology Dispensary #4, Saint Petersburg
  - LLC International Medical Centre "SOGAZ", Saint Petersburg
- South Africa (5):
  - Cape Trial Centre, Cape Town, W. Cape
  - Paarl Medical Centre, Paarl, W. Cape
  - Clinika, Port Elizabeth, E. Cape
  - Dey Clinic, Pretoria, Gauteng
  - Vereeniging Medi-Clinic, Vereeniging, Free State
- Ukraine (5):
  - Reg. Clinic Psych. Hosp., Dept 11, DNMU n.a.M. Gorkiy, Donetsk
  - Odesa Regional Psychoneurological Dispensary, Odesa
  - Reg. Ci.Ps.H.n.a.O.F.Maltsev, Fem.Ac.Gen.Ps. D.5B,HESIU UM, Poltava
  - CRI"Cl. Psych.Hosp.#1, Fem Psych.Dept.#2, Male Psych.Dept.#1, Simferopol
  - Reg. Psych. Hosp. n.a. O.Yuschenko, Dept. #21, VNMUn.a.M. Pirog, Vinnitsia

REFERENCES:
- [Result] Loebel A, Cucchiaro J, Silva R, Kroger H, Sarma K, Xu J, Calabrese JR. Lurasidone as adjunctive therapy with lithium or valproate for the treatment of bipolar I depression: a randomized, double-blind, placebo-controlled study. Am J Psychiatry. 2014 Feb;171(2):169-77. doi: 10.1176/appi.ajp.2013.13070985. PMID 24170221
- [Derived] Tocco M, Mao Y. Efficacy and Safety of Adding Lurasidone to Ongoing Therapy With Lithium or Valproate for the Treatment of an Acute Bipolar Depressive Episode: A Post Hoc Analysis of 2 Placebo-Controlled Trials. J Clin Psychopharmacol. 2024 Jul-Aug 01;44(4):345-352. doi: 10.1097/JCP.0000000000001850. Epub 2024 Apr 19. PMID 38639433
- [Derived] Goldberg JF, Siu C, Tocco M, Pikalov A, Loebel A. The Effect of Lurasidone on Anxiety Symptoms in Patients With Bipolar Depression: A Post Hoc Analysis. J Clin Psychiatry. 2023 Jun 7;84(4):22m14732. doi: 10.4088/JCP.22m14732. PMID 37339360
- [Derived] Sajatovic M, Forester BP, Tsai J, Kroger H, Pikalov A, Cucchiaro J, Loebel A. Efficacy of Lurasidone in Adults Aged 55 Years and Older With Bipolar Depression: Post Hoc Analysis of 2 Double-Blind, Placebo-Controlled Studies. J Clin Psychiatry. 2016 Oct;77(10):e1324-e1331. doi: 10.4088/JCP.15m10261. PMID 27529375
- [Derived] Rajagopalan K, Bacci ED, Ng-Mak D, Wyrwich K, Pikalov A, Loebel A. Effects on health-related quality of life in patients treated with lurasidone for bipolar depression: results from two placebo controlled bipolar depression trials. BMC Psychiatry. 2016 May 23;16:157. doi: 10.1186/s12888-016-0865-y. PMID 27215976
- [Derived] Chapel S, Chiu YY, Hsu J, Cucchiaro J, Loebel A. Lurasidone Dose Response in Bipolar Depression: A Population Dose-response Analysis. Clin Ther. 2016 Jan 1;38(1):4-15. doi: 10.1016/j.clinthera.2015.11.013. Epub 2015 Dec 22. PMID 26730454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5/11/2009 - 1/9/2012
Groups:
- Lurasidone: lurasidone + (lithium or divalproex) : lurasidone 20 mg/day for Days 1-2-3, 40 mg/day for Days 4-5-6, and 60 mg/day on Day 7.
- Placebo: Placebo + (lithium or divalproex) : 20 mg/day for Days 1-2-3, 40 mg/day for Days 4-5-6, and 60 mg/day on Day 7
Period: Overall Study
Arm/Group | Lurasidone | Placebo
Started | 183 | 165
Completed | 143 | 136
Not Completed | 40 | 29

BASELINE CHARACTERISTICS:
Population: Data for full analysis set is provided (intent-to-treat population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone | Placebo | Total
Number analyzed (Participants) | 179 | 161 | 340
Age, Categorical [Count of Participants; unit: Participants] — Data for full analysis set is provided.
  Participants
    <=18 years | 0 | 1 | 1
    Between 18 and 65 years | 178 | 155 | 333
    >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] — Data for full analysis set is provided.
  years | 41.0 (11.53) | 42.6 (11.75) | 41.7 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 76 | 162
  Male | 93 | 85 | 178
Region of Enrollment [Number; unit: participants]
  France | 8 | 8 | 16
  United States | 58 | 52 | 110
  Czech Republic | 27 | 21 | 48
  Poland | 9 | 6 | 15
  Ukraine | 11 | 12 | 23
  Romania | 2 | 3 | 5
  South Africa | 10 | 8 | 18
  Russian Federation | 9 | 10 | 19
  Germany | 2 | 4 | 6
  India | 43 | 37 | 80

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Endpoint (Week 6)
Description: MADRS total score ranges from a minimum of 0 to a maximum of 60. Lower values represent a better score, higher values represent a worse score. Similarly, greater negative change from baseline represents improvement, and positive changes from baseline represent worsening.
Time Frame: Baseline, Week 6
Population: Full analysis set (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 179 | 161
units on a scale | -17.1 (0.87) | -13.5 (0.91)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; Mean Difference (Final Values) = -3.6, Standard Error of Mean 1.25

2. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 6) in: Clinical Global Impression Bipolar Version, Severity of Illness (CGI-BP-S) Score (Depression)
Description: CGI-EP-S depression score ranges from a minimum of 0 to a maximum of 7. Lower values represent a better score, higher values represent a worse score. Similarly, greater negative change from baseline represents improvement, and positive changes from baseline represent worsening.
Time Frame: Baseline Week 6
Population: Full analyis set (intent-to-treat population)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 179 | 161
units on a scale | -1.96 (0.104) | -1.51 (0.109)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mean Difference (Final Values) = -0.44, Standard Error of Mean 0.150

3. Secondary Outcome: Mean Change From Baseline to Endpoint (Week 6) in: Sheehan Disability Scale (SDS) Total Score
Description: STS total score ranges from a minimum of 0 to a maximum of 30. Lower values represent a better score, higher values represent a worse score. Similarly, greater negative change from baseline represents improvement, and positive changes from baseline represent worsening.
Time Frame: Baselin Week 6
Population: Full analysis set (intent-to-treat population)
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 179 | 161
units on a scale | -9.5 (0.78) | -7.0 (0.81)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA; Mean Difference (Final Values) = -2.6, Standard Error of Mean 1.01

ADVERSE EVENTS:
Time Frame: Adverse event reporting begins at time of informed consent signature and continues until patient discontinuatiion - 6 Weeks
Description: Number of participants at risk is the Safety Analysis Set (all randomized subjects exposed to at least one dose of study medicaton).
Arm/Group | Lurasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 2/183 | 2/163
Other Adverse Events (participants affected / at risk) | 73/183 | 51/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=183) | Placebo (N=163)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone (N=183) | Placebo (N=163)
Nausea (Gastrointestinal disorders) | 32 (44) | 18 (24)
Headache (Nervous system disorders) | 19 (30) | 20 (29)
Somnolence (Nervous system disorders) | 17 (17) | 7 (9)
Tremor (Nervous system disorders) | 15 (17) | 7 (8)
Akathisia (Nervous system disorders) | 14 (18) | 7 (10)
Insomnia (Psychiatric disorders) | 13 (21) | 9 (11)
Diarrhea (Gastrointestinal disorders) | 8 (10) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.